CLINICAL TRIAL: NCT01216904
Title: Nicotine Treatment of Impulsivity in Parkinson's Disease: A Pilot Study
Brief Title: Nicotine Treatment of Impulsivity in Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: Parkinson's Disease Foundation (Other); The Parkinson Study Group (Network)
Responsible Party: Principal Investigator, James BOYD MD, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PSG PDF MCRA 07012010
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo patch (Placebo Comparator)
  Interventions: Drug: placebo
- Nicotine patch (Active Comparator)
  Interventions: Drug: nicotine patch

INTERVENTIONS:
Drug: nicotine patch — 7 mg patches to be worn for 16 hours per day
  Other Names: Nicoderm patches
  Arms: Nicotine patch
Drug: placebo — placebo patch to be worn 16 hours per day
  Arms: Placebo patch

SUMMARY:
The specific aims of this study are to examine whether treatment with transdermal nicotine improves computer-based laboratory and clinical measures of impulsive and compulsive behaviors in Parkinson's Disease subjects who have recently experienced an impulse control disorder.

DETAILED DESCRIPTION:
In recent years, a group of behavior changes collectively called Impulse Control Disorders (ICDs) have been identified in Parkinson's Disease (PD). ICDs have a broad range of possible symptoms such as compulsive gambling, shopping, hypersexual behavior, overeating; spending excessive amounts of time on hobbies, tasks, or other organized activities; walking or driving without a goal or purpose; hoarding or overuse of PD medications. It is estimated that as many as 30% of people with PD experience ICDs during the course of their condition. ICDs are believed to occur due to effects of dopamine enhancing medications in areas of the brain which regulate behavior (rather than their intended target areas that regulate movement).

A reduction or discontinuation of PD medications can be helpful in reducing ICDs. Unfortunately reduction in medication is often impractical or not possible because people with PD rely on these medications to improve their movement symptoms. There are currently no scientifically proven treatments for ICDs except for PD medication reductions.

Acetylcholine is a chemical in the brain which works to regulate the effects of dopamine. It has been known for many years that nicotine imitates many of the actions of acetylcholine. In preliminary studies, nicotine has been shown to reduce impulsive behavior in Attention Deficit Hyperactivity Disorder. By administering nicotine across the skin using a patch, we hope to better understand whether nicotine may act to improve impulse control disorders in PD without needing to reduce or stop PD medications. Several studies have shown that nicotine is tolerated well by people with PD, and does not appear to worsen motor/movement symptoms. The amount of nicotine in each patch used in this study is the same as patches that are used in people who are trying to quit smoking.

In this pilot within-subject crossover placebo-controlled study, subjects with a diagnosis of Parkinson's Disease who have recently experiencing an impulse control disorder will be enrolled. Subjects will randomized to one of two treatment groups. During the first portion of the study, the first treatment group will receive transdermal nicotine (nicotine by skin patch) and the second treatment group will receive an identical placebo patch which does not contain any nicotine. Over the course of the study, each of the two groups will switch to receive whichever treatment they were not initially receiving (for example-the first treatment group will later receive the placebo patch and the second treatment group will later receive the nicotine patch). Each treatment group will receive the nicotine patch or placebo patch for an equal number of weeks, but at different times during the study. Clinical and laboratory computer based measurements of impulsive and compulsive behaviors, memory testing, sleep quality/ sleepiness, and Parkinson's disease symptoms will be assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of idiopathic Parkinson's Disease based on movement disorders specialist assessment using the National Institute of Neurological disorders and Stroke (NINDS) criteria 17;
* demonstrated response to L-¬DOPA and/or dopamine agonists;
* Hoehn and Yahr19 stage 1 - 3 motor disability in the "on" medication state;
* stable PD and non-PD medications for at least 1 month prior to baseline;
* positive QUIP screening and confirmatory interview for current or prior ICD symptoms 36;
* Montreal Cognitive Assessment score > 24;
* impaired impulsive and/or compulsive responding compared to norms on Stop Signal Task and/or Set-Shifting Task
* Global Deterioration Scale score24 of 1-2;
* Adequate visual and auditory acuity for neuropsychological testing;
* good general health with no additional diseases expected to interfere with the study;
* normal laboratory tests and ECG;
* female participants must be non-breastfeeding, post-menopausal or have been surgically sterilized or have a negative urine pregnancy test at screening and baseline visits with an acceptable form of contraception being used (see drug safety section for details on acceptable contraception);
* Subjects will be taking no centrally active or anti or pro-cholinergic drugs;
* non¬smokers, defined as no cigarettes in the last 6 months

Exclusion Criteria:

* severe motor fluctuations;
* prior DBS surgery;
* Any significant systemic illness or unstable medical condition including serious heart disease, severe asthma, severe or active ulcer disease, active thyroid disease, pyloric stenosis epilepsy, or allergies to nicotine;
* clinically significant laboratory test abnormalities on the battery of screening tests (hematology, chemistry, urinalysis, ECG);
* uncontrolled hypertension (systolic BP> 170 or diastolic BP> 100);
* Any current significant or unstable depression, anxiety, or psychosis
* history of obsessive-compulsive disorder
* use of any investigational drugs within 30 days or 5 half-¬lives, whichever is longer, prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Stop Signal task | 15 minutes
  The Stop Signal Task is best described as a laboratory measure of inhibitory control. The task itself requires quick execution of a thought or action, and the occasional inhibition of this behavior. On the computerized task subjects are asked to respond as fast as they can to symbols (ex. letters) presented on a computer screen.

SECONDARY OUTCOMES:
Set shifting task | 12-20 minutes
  It has been considered a measure of executive function because of its reported sensitivity to frontal lobe dysfunction. As such, the WCST allows the clinician to assess the following "frontal" lobe functions: strategic planning, organized searching, utilizing environmental feedback to shift cognitive sets, directing behavior toward achieving a goal, and modulating impulsive responding.

CONTACTS AND LOCATIONS:
Overall Officials: James Boyd, MD, Principal Investigator — UVM/FAHC
Locations (1):
- Fletcher Allen Health Care/UVM, Burlington, Vermont, United States